CLINICAL TRIAL: NCT07323381
Title: A Multicenter, Randomized, Parallel-group Clinical Study on the Effects of Henagliflozin Proline Tablets and Metformin Sustained-release Tablets on Body Composition in Geriatric Patients With Newly Diagnosed Type 2 Diabetes Mellitus
Brief Title: Effects of Henagliflozin Proline and Metformin XR on Body Composition in Geriatric Patients With Newly Diagnosed T2DM
Acronym: HABIT-GEMs
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bin Lu (Other)
Collaborators: Shanxi Provincial People's Hospital (Other Government); Zhongnan Hospital (Other); Second Affiliated Hospital of Soochow University (Other); The Second Affiliated Hospital of Shandong First Medical University (Other); Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor-Investigator, Bin Lu, Principal Investigator, Director, Clinical Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025K268
Record Dates: First submitted 2025-12-04; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Diabetes Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Henagliflozin Proline Tablets treatment group (Experimental): Drug: Henagliflozin Proline Tablets treatment Start with a once-daily dose of either Henagliflozin Proline Tablets (5mg) ,with a potential dose adjustment at Week 12.
  Interventions: Drug: Henagliflozin Proline Tablets treatment
- Metformin Sustained-release tablets treatment group (Experimental): Start with a once-daily dose of either Metformin XR (1000mg), with a potential dose adjustment at Week 12.
  Interventions: Drug: Metformin XR treatment

INTERVENTIONS:
Drug: Henagliflozin Proline Tablets treatment — Start with a once-daily dose of either Henagliflozin Proline Tablets (5mg) , with a potential dose adjustment at Week 12.
  Arms: Henagliflozin Proline Tablets treatment group
Drug: Metformin XR treatment — Start with a once-daily dose of either Metformin XR (1000mg), with a potential dose adjustment at Week 12.
  Arms: Metformin Sustained-release tablets treatment group

SUMMARY:
The goal of this clinical trial is to compare the effects of Henagliflozin Proline Tablets versus Metformin Extended-Release on body composition in elderly, drug-naïve patients with Type 2 Diabetes. The main questions it aims to answer are:

The effect of each treatment on the change in body composition, as measured by Appendicular Skeletal Muscle Index (ASMI), from baseline to 24 weeks.

The effect of each treatment on the change in HbA1c from baseline to 24 weeks. The comparative safety profile and other efficacy measures (e.g. fasting plasma glucose and additional body composition parameters) between the two treatments.

Researchers will compare the Henagliflozin Proline treatment group to the Metformin Extended-Release treatment group to evaluate potential differences in changes in muscle mass and metabolic parameters.

Participants will:

Be randomly assigned to one of the two treatment groups. Attend multiple clinic visits and telephone follow-ups over a 28-week period.

At clinic visits, undergo procedures including:

Physical examinations (height, weight, blood pressure, circumferences). Body composition analysis using bioelectrical impedance analysis (BIA). Physical function tests (handgrip strength, 5-times sit-to-stand test, 6-meter walk speed).

Blood and urine tests for efficacy and safety biomarkers. Dietary recording and exercise guidance. Start with a once-daily dose of either Henagliflozin Proline (5 mg) or Metformin XR (1000 mg), with a potential dose adjustment at Week 12.

ELIGIBILITY:
Inclusion Criteria:

Voluntarily sign the informed consent form, be able to understand the procedures and methods of this study, and be willing to strictly comply with the clinical trial protocol to complete the study.

Aged between 60 and 85 years (inclusive) at the time of screening, regardless of gender.

Diagnosed with Type 2 Diabetes Mellitus according to WHO criteria, and not having used any glucose-lowering medications in the recent 3 months.

7.0% ≤ HbA1c ≤ 11.0% and Fasting Plasma Glucose ≤ 15 mmol/L. Body fat percentage: ≥25% for males, ≥30% for females.

Exclusion Criteria:

Known or suspected allergy to metformin, SGLT2 inhibitors, or excipients of the investigational product.

History of Type 1 Diabetes or other forms of insulin-dependent diabetes. Acute metabolic complications within the past 6 months, such as ketoacidosis, lactic acidosis, or hyperosmolar coma.

History of severe or recurrent hypoglycemic episodes. Presence of diabetes insipidus. Unstable thyroid function with treatment doses not stabilized within the past 3 months.

History of cardiovascular events within the past 6 months. Patients with uncontrolled hypertension or hypotension. Presence of clinical symptoms or recurrent urinary tract infections or genital infections.

History of osteoporosis, hematological diseases, malignancy, significant gastrointestinal disorders, fluid retention states, hypovolemia, or uncontrolled psychiatric disorders.

Systemic corticosteroid therapy for more than 7 days within the past 3 months. History of bariatric surgery within the past 12 months, use of weight-control medications within the past 3 months, or current participation in a weight-loss program not in the maintenance phase.

Gastrointestinal surgery that affects absorption within the past 3 months; long-term use of medications directly affecting gastrointestinal motility; or acute stress conditions such as surgery, infection, or hospitalization within the past 3 months.

Participation in any other drug clinical trial within the past 3 months. ALT or AST levels > 3 times the upper limit of normal; Hemoglobin ≤ 100 g/L; Renal impairment, defined as eGFR < 45 mL/min/1.73 m²; Fasting triglycerides ≥ 5.64 mmol/L.

History of diabetic retinopathy. Significantly abnormal 12-lead ECG. Any other condition deemed by the investigator as unsuitable for the subject's participation in this study.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in body composition (Appendicular Skeletal Muscle mass / Height² kg/m² weight in kilograms, height in meters) from baseline to Week 24. | from baseline to Week 24
  Appendicular skeletal muscle mass index (ASMI, kg/m²) will be derived from bioelectrical impedance analysis (BIA) measurements. ASMI is calculated as appendicular skeletal muscle mass (ASM, kg) divided by height squared (m²). ASM will be estimated using a BIA device. Measurements will be performed at baseline (V0) and at week 24 (V6), following a standardised protocol that includes ≥4 hours of fasting. The ASM value will be generated by the device's integrated software.

SECONDARY OUTCOMES:
Change in appendicular skeletal muscle mass relative to body weight (ASM/BW) from baseline to Week 24. | from baseline to Week 24
  ASM/BW is a unitless ratio (kg/kg) of appendicular skeletal muscle mass to total body weight. Both components will be measured using a bioelectrical impedance analysis (BIA) device, following a standardized protocol that includes participant fasting and rest prior to measurement. The ratio will be calculated from the raw BIA estimates of appendicular skeletal muscle mass and total body weight generated by the device software.
Change in HbA1c from baseline to Week 24. | from baseline to Week 24
  HbA1c: Assessed from venous blood samples collected after a required fast. Analysis will be performed using a standardized, high-performance liquid chromatography (HPLC) method in a certified central laboratory at Baseline and Week 24.
Change in body fat percentage from baseline to Week 24. | from baseline to Week 24
  Body fat percentage (BF%) is a unitless index calculated as estimated total body fat mass (in kg) divided by estimated total body weight (in kg), multiplied by 100%. Both fat mass and total body weight will be estimated by a bioelectrical impedance analysis (BIA) device, following a standardised pre-measurement protocol which includes fasting and rest.